CLINICAL TRIAL: NCT02362256
Title: The Comparison of Stress Response to Rapid Opioid Detoxification Applying Different Methods of Opioid Antagonism With Naltrexone and Sedation
Brief Title: The Comparison of Stress Response to Rapid Opioid Detoxification Applying Different Methods of Opioid Antagonism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Robertas Badaras, MD Robertas Badaras, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 158200-01-443-124
Record Dates: First submitted 2015-01-18; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Opiate Addiction
Keywords: Opioid detoxification; Opioid antagonist induction; Conscious sedation
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; vivitrol; Clonidine; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Opioid antagonist induction. Day 4. Duration 12-16 hours.
  Naltrexone gradual increase from 50 µg p/o to a total dose of 12,5 mg according to a predefined protocol:
  1. st hour 50 µg
  2. nd hour 50 µg
  3. rd hour 100 µg
  4. th hour 100 µg
  5. th hour 200 µg
  6. th hour 400 µg
  7. th hour 800 µg
  8. th hour 1600 µg
  9. th hour 3200 µg
  10. th hour 6000 µg
  Correction of symptoms for opioid abstinence:
  Clonidine 150 µg p/o every 4 hours (Day 3 and Day 4) Lorazepam 5 mg p/o every 4 hours (Day 3 and Day 4), Lorazepam 2,5 mg po every 4 hours (Day 5, Day 6)
  Interventions: Drug: Naltrexone; Drug: Clonidine; Drug: Lorazepam
- Control (Active Comparator): Opioid antagonist induction. Day 4. Duration 12-16 hours. Naltrexone single dose 12,5 mg p/o
  Correction of symptoms for opioid abstinence:
  Clonidine 150 µg p/o every 4 hours (Day 3 and Day 4) Lorazepam 5 mg p/o every 4 hours (Day 3 and Day 4), Lorazepam 2,5 mg po every 4 hours (Day 5, Day 6)
  Interventions: Drug: Naltrexone; Drug: Clonidine; Drug: Lorazepam

INTERVENTIONS:
Drug: Naltrexone
  Other Names: Vivitrol; Revia
Drug: Clonidine
  Other Names: Catapres; Kapvay
Drug: Lorazepam
  Other Names: Ativan

SUMMARY:
The aim of this study is to investigate which method of naltrexone induction during rapid opioid detoxification causes stronger stress response and has a higher influence on opioid abstinence caused by opioid induction.

DETAILED DESCRIPTION:
Study enrolls opiate addicted patients who are motivated for a long term treatment and full opiate abstinence. Patient is offered to take part in a study. Information is provided regarding protocol, aim and course of study. Patients who are eligible and consent for study commit to follow the pre-study recommendations.

Study consists of:

Primary assessment - information about study. Assessment of patient according to predefined criteria. Consent form. Allocation of the treatment date.

Stabilization - Buprenorphine. Assessment according to SOWS and OWS. Total amount of buprenorphine is recorded.

Repeated evaluation - patient after successful stabilization course undergoes urine test for psychotropic substances, blood alcohol level is recorded. If any test is positive patient is not enrolled to study.

Correction of opioid withdrawal symptoms - all of the patients receive medicines for opioid detoxification, infusion therapy in predefined doses.

Antagonist induction - patients receive opioid antagonist (incremental or standard dose). Withdrawal symptoms are assessed and correction with lorazepam is given if needed.

Data collection - data is recorded (demographic, epidemiological, vital signs, opioid withdrawal symptoms, levels of hormones, metabolites, electrolytes).

ELIGIBILITY:
Inclusion Criteria:

* Opiate addiction
* Use of short-acting opiate (morphine or heroine)
* Age > 18 years
* Length of opiate addiction > 1 year
* Patient can make a decision for detoxification and has a capacity to consent for procedure
* Written consent for procedure

Exclusion Criteria:

* Polyvalent addiction
* Pregnancy or breast feeding
* Cardiovascular pathology
* Acute or chronic kidney disease
* Decompensated liver pathology (jaundice, ascites, hepatic encephalopathy)
* Infective complications of opiate addiction (pneumonia, phlegmon, abscess, thombophlebitis, sepsis)
* Malnutrition (Nutritional risk screening 2002 score ≥3)
* Diabetes mellitus
* Previous history of psychosis
* Glasgow coma scale < 15
* Abdominal surgical intervention during last 30 days
* Cumulative buprenorphine dose for stabilization < 8 mg
* Positive test for psychoactive substances during treatment
* Refusal to participate in study at any point of it

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cortisol levels | 2 days
  Cortisol levels were assessed 4 times starting on intervention day (1 hour before intervention, 1, 5 and 23 hours post-intervention)
Adrenocorticotropic hormone (ACTH) levels | 2 days
  Cortisol levels were assessed 4 times starting on intervention day (1 hour before intervention, 1, 5 and 23 hours post-intervention)

SECONDARY OUTCOMES:
Stress response levels according to heart rate | 4 days
  Heart rate measurements were taken 4 times a day
Stress response levels according to respiratory rate | 4 days
  Respiratory rate measurements were taken 4 times a day
Stress response levels according to blood pressure | 4 days
  Blood pressure measurements were taken 4 times a day
Changes of potassium concentration due to stress response | 4 days
  Blood samples were taken 3 times a day
Changes of sodium concentration due to stress response | 4 days
  Blood samples were taken 3 times a day
Changes of chloride concentration due to stress response | 4 days
  Blood samples were taken 3 times a day
Changes of magnesium concentration due to stress response | 4 days
  Blood samples were taken 3 times a day
Changes of glucose concentration due to stress response | 4 days
  Blood samples were taken 3 times a day
Subjective Opiate Withdrawal Scale (SOWS) | 4 days
  Patients were assessed with to SOWS 4 times a day
Objective Opiate Withdrawal Scale (OOWS) | 4 days
  Patients were assessed with to OOWS 4 times a day

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTAS BADARAS, MD, Principal Investigator — Vilnius University Clinic of Anaesthesiology and Intensive Care; JUOZAS IVASKEVICIUS, PROFESSOR, Study Director — Vilnius University Clinic of Anaesthesiology and Intensive Care
Locations (1):
- Republic Vilnius University Hospital, Vilnius, Vilnius County, Lithuania